CLINICAL TRIAL: NCT03158610
Title: Biological-guided Metronomic Chemotherapy as Maintenance Strategy in Responders After Induction Therapy in Metastatic Colorectal Cancer
Brief Title: Biological-guided Metronomic Chemotherapy as Maintenance Strategy in Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Difficult to enrollment patient
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhang, Deputy-chief of Department of Oncology, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIG-MOON
Record Dates: First submitted 2017-05-15; First posted 2017-05-18 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capecitabine metronomic chemotherapy (Experimental): Capecitabine 500mg/m2 bid po qd
  Interventions: Drug: Capecitabine
- Capecitabine standard dosage chemotherapy (Active Comparator): Capecitabine 1000mg/m2 bid po d1-d14,q3w
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Oral fluorouracil
  Other Names: Xeloda

SUMMARY:
Based upon biological behavior, those mCRC patients who respond well (SD, PR or CR according to RECIST Criteria) after 16-18 weeks of standard doublet chemotherapy as induction may enrolled into this study, randomly divided into capecitabine metronomic group or standard dosage group. The duration of disease control after randomization(PFS2) and progression free survival from enrollment (PFS1) are primary endpoints. Meanwhile, the overall survival, safety and quality of life are secondary endpoints. Exploratory markers involving angiogenesis (serum VEGF, PDGF, Tie-1 and Tie2, etc) and immune function (CD clusters, serum tumor mutation burden(TMB), etc), are conducted via liquid biopsy.

DETAILED DESCRIPTION:
This study is try to evaluate the effect of capecitabine metronomic chemotherapy as maintenance treatment, which compare to capecitabine conventional chemotherapy, who have responded to 16-18 months first-line chemotherapy in metastatic colorectal cancer (mCRC). The maintenance treatments are continued until disease progression or severe toxicity. The aim of this study is to demonstrate that capecitabine metronomic chemotherapy is non-inferior to capecitabine conventional chemotherapy. Furthermore, exploratory markers involving angiogenesis (serum VEGF, PDGF, Tie-1 and Tie2, etc) and immune function (CD clusters, serum tumor mutation burden(TMB), etc), are conducted via liquid biopsy.

ELIGIBILITY:
Before the start of induction therapy:

Inclusion Criteria:

* Histological proof of colorectal cancer (in case of a single metastasis, histological or cytological proof of this lesion should be obtained);
* Distant metastases which are unresectable (patients with only local recurrence are not eligible);
* Measurable disease (> 1 cm on spiral CT scan or > 2 cm on chest X-ray; liver ultrasound is not allowed). Serum CEA may not be used as a parameter for disease evaluation;

Exclusion criteria

* Prior adjuvant treatment for stage II/III colorectal cancer ending within 6 months before the start of induction treatment
* Any prior adjuvant treatment after resection of distant metastases
* Previous systemic treatment for advanced disease

At randomisation:

Inclusion criteria:

* WHO performance status 0-1 (Karnofsky PS > 70%);
* Disease evaluation with proven SD, PR or CR according to RECIST after first-line induction treatment;
* Laboratory values obtained ≤ 2 weeks prior to randomisation: adequate bone marrow function (Hb > 6.0 mmol/L, absolute neutrophil count > 1.5 x 109/L, platelets > 100 x 109/L), renal function (serum creatinine ≤ 1.5x ULN and creatinine clearance, Cockroft formula, > 30 ml/min), liver function (serum bilirubin ≤ 2 x ULN, serum transaminases ≤ 3 x ULN without presence of liver metastases or ≤ 5x ULN with presence of liver metastases);
* Life expectancy > 12 weeks;
* Age: 18-75 years;
* Negative pregnancy test in women with childbearing potential;
* Expected adequacy of follow-up;
* Institutional Review Board approval;
* Written informed consent Exclusion criteria
* Chronic active infection;
* Any other concurrent severe or uncontrolled disease preventing the safe administration of study drugs;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival 1 (PFS1) | 10 months
  from enrollment to progression
Progression Free Survival 2 (PFS2) | 4 months
  from randomization to progression

SECONDARY OUTCOMES:
Overall Survival (OS) | 20 months
  from signing informed consent to death
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 20 months
  drug related toxicity from signing informed consent to death
Number of participants with quality of life (QoL) as assessed by CTCAE v4.0 | 20 months
  QoL from signing informed consent to death

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD & Ph. D, Principal Investigator — Ruijin Hospital
Locations (1):
- Department of Oncology, Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kareva I, Waxman DJ, Lakka Klement G. Metronomic chemotherapy: an attractive alternative to maximum tolerated dose therapy that can activate anti-tumor immunity and minimize therapeutic resistance. Cancer Lett. 2015 Mar 28;358(2):100-106. doi: 10.1016/j.canlet.2014.12.039. Epub 2014 Dec 23. PMID 25541061
- [Background] Tournigand C, Cervantes A, Figer A, Lledo G, Flesch M, Buyse M, Mineur L, Carola E, Etienne PL, Rivera F, Chirivella I, Perez-Staub N, Louvet C, Andre T, Tabah-Fisch I, de Gramont A. OPTIMOX1: a randomized study of FOLFOX4 or FOLFOX7 with oxaliplatin in a stop-and-Go fashion in advanced colorectal cancer--a GERCOR study. J Clin Oncol. 2006 Jan 20;24(3):394-400. doi: 10.1200/JCO.2005.03.0106. PMID 16421419
- [Background] Andre T, Tournigand C, Mineur L, Fellague-Chebra R, Flesch M, Mabro M, Hebbar M, Postel Vinay S, Bidard FC, Louvet C, de Gramont A. Phase II study of an optimized 5-fluorouracil-oxaliplatin strategy (OPTIMOX2) with celecoxib in metastatic colorectal cancer: a GERCOR study. Ann Oncol. 2007 Jan;18(1):77-81. doi: 10.1093/annonc/mdl336. Epub 2006 Oct 9. PMID 17030548
- [Background] Simkens LH, van Tinteren H, May A, ten Tije AJ, Creemers GJ, Loosveld OJ, de Jongh FE, Erdkamp FL, Erjavec Z, van der Torren AM, Tol J, Braun HJ, Nieboer P, van der Hoeven JJ, Haasjes JG, Jansen RL, Wals J, Cats A, Derleyn VA, Honkoop AH, Mol L, Punt CJ, Koopman M. Maintenance treatment with capecitabine and bevacizumab in metastatic colorectal cancer (CAIRO3): a phase 3 randomised controlled trial of the Dutch Colorectal Cancer Group. Lancet. 2015 May 9;385(9980):1843-52. doi: 10.1016/S0140-6736(14)62004-3. Epub 2015 Apr 7. PMID 25862517
- [Derived] Shi M, Ma T, Xi W, Jiang J, Wu J, Zhou C, Yang C, Zhu Z, Zhang J. A study of capecitabine metronomic chemotherapy is non-inferior to conventional chemotherapy as maintenance strategy in responders after induction therapy in metastatic colorectal cancer. Trials. 2020 Mar 6;21(1):249. doi: 10.1186/s13063-020-4194-6. PMID 32143730